CLINICAL TRIAL: NCT00734825
Title: Emergency Department CT Scanning for Appendicitis: IV Contrast vs. IV and Oral Contrast
Brief Title: Emergency Department CT Scanning for Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Andrew Kepner, MD / Medical Director, WellSpan Health Simulation Center, WellSpan HEalth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0607012
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Appendicitis
Keywords: Appendicitis; IV Contrast; Oral Contrast; CT scan
MeSH Terms: conditions — Appendicitis | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): IV contrast
  Interventions: Other: Omnipaque
- 2 (Active Comparator): IV contrast and oral contrast
  Interventions: Other: Omnipaque

INTERVENTIONS:
Other: Omnipaque — oral contrast for CT scan

SUMMARY:
The purpose of this study is to compare IV contrast only vs. IV and oral contrast Computed Tomography (CT) for the diagnosis of acute appendicitis in adult patients in our emergency department. A secondary purpose will be to design a specific CT for appendicitis protocol at our institution at the conclusion of this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older who present to the York Hospital Emergency Department with signs and symptoms suggestive of acute appendicitis, but in whom the diagnosis remains unclear as determined by an attending emergency physician or consulting surgeon and in which a CT scan is needed to further assist in the diagnosis

Exclusion Criteria:

* pregnant patients
* patients with known IV dye or oral contrast allergy
* patients in whom acute appendicitis is not the primary diagnosis
* patients with renal insufficiency that may have significant adverse effect from IV dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
sensitivity of IV contrast alone for a computed tomography scan for the diagnosis of appendicitis in the adult Emergency Department patient. | immediate reading + blinded reading within 48 hours

SECONDARY OUTCOMES:
If IV contrast alone for CT scan is sensitive for the diagnosis of appendicitis in the adult Emergency department patient | immediate reading and blinded reading within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kepner, MD, Principal Investigator — WellSpan Health

REFERENCES:
- [Derived] Kepner AM, Bacasnot JV, Stahlman BA. Intravenous contrast alone vs intravenous and oral contrast computed tomography for the diagnosis of appendicitis in adult ED patients. Am J Emerg Med. 2012 Nov;30(9):1765-73. doi: 10.1016/j.ajem.2012.02.011. Epub 2012 May 23. PMID 22633722